CLINICAL TRIAL: NCT04749030
Title: Faecal Microbiota Transplantation for Patients With Diabetes Mellitus Type 1 and Severe Gastrointestinal Neuropathy: a Randomised, Double-blinded Safety and Pilot-efficacy Study
Brief Title: Faecal Microbiota Transplantation for Patients With Diabetes Mellitus Type 1 and Severe Gastrointestinal Neuropathy
Acronym: Fadigas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Fadigas
Record Dates: First submitted 2021-02-01; First posted 2021-02-10 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2022-05

CONDITIONS: Faecal Microbiota Transplantation (FMT); Diabetes Mellitus, Type 1; Gastrointestinal Neuropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Fecal Microbiota Transplantation; Capsules

STUDY DESIGN:
Intervention Model Description: The study is a 8-week, randomised, double-blinded, placebo-controlled pilot trial of oral FMT versus placebo in patients with DM1 and severe GI neuropathy. The intervention period consists of a first 4 weeks where patients receive either FMT or placebo and a second 4 weeks where all patients receive FMT. The patients will undergo the investigations before and after each 4-week period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Faecal microbiota transplantation (FMT) (Other): Donor faeces is obtained from thoroughly screened healthy blood donors and processed in compliance with the European Tissue and Cells Directive.
  Interventions: Other: Faecal microbiota transplantation (FMT) capsules
- Placebo (Placebo Comparator): Placebo capsules will be identical in terms of visual appearance, weight, and vials and number
  Interventions: Other: Placebo capsules

INTERVENTIONS:
Other: Faecal microbiota transplantation (FMT) capsules — The faeces is minimally processed through a series of centrifugation steps and dispensed into double-coated, acid resistant enterocapsules. A single treatment includes approximately 22 capsules (~50 grams of original donor faeces).
  Arms: Faecal microbiota transplantation (FMT)
Other: Placebo capsules — The placebo capsules are produced from a suspension of 50% glycerol, 40% sterile saline and 10% food coloring in enterocapusles
  Arms: Placebo

SUMMARY:
A randomised, double-blinded and placebo-controlled intervention study. The study aim to evaluate the feasibility, safety and pilot-efficacy of faecal microbiota transplantation as a treatment of severe gastrointestinal neuropathy in patients with diabetes mellitus type 1.

DETAILED DESCRIPTION:
Diabetes type 1 may cause damage to nerve cells in the gut causing neuropathy that leads to changes in gastric and intestinal motility. This change predisposes to an abnormal amounts and composition of bacteria in the gut, probably leading to uncontrollable diarrhea and severely impaired quality of life. Transferal of intestinal microbiota from a healthy donor to a patient is called faecal microbiota transplantation (FMT). FMT may potentially change the bacteria in the gut and reduce gastrointestinal symptoms. However, FMT may also have potential side effects, especially in persons with autonomic neuropathy and delayed transit through the gut.

ELIGIBILITY:
Inclusion Criteria:

Adult (≥ 18 years old), male or female patients with DM1 for at least 5 years and average of or above 40 points in the questionnaire: Gastrointestinal syndrome rating scale - irritable bowel syndrome version (GSRS-IBS).

Exclusion Criteria:

* Inability to understand Danish or the trial procedures
* Known or anticipated pregnancy
* Known severe renal insufficiency
* Antibiotic use in the prior 4 weeks
* Treatment with morphine
* Ongoing infection with Clostridioides difficile or pathogenic intestinal bacteria or parasites
* Known gastrointestinal disease or GI infection
* Patients diagnosed with intestinal stricture
* Patients with other known disorder that can cause gastroparesis
* Patients with planned MR scan within 4 weeks
* Patients with pacemaker/ICD
* Previous abdominal surgery
* Changes in medicine that affects the GI tract in the prior 4 weeks

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Number of adverse events of severity grade 2 or more assessed by CTCAE v5.0 during the first week after first intervention (FMT or placebo). | One week after the first intervention
  Patient-reported measures from the schedule of side effects and telephone call 1 week after each intervention.

SECONDARY OUTCOMES:
Patient-reported outcomes obtained from the bowel habit diary. | Each patient fills out the diary every day for one week at baseline, for one week starting at each day of the two interventions and for one week at the long term follow-up at week 26
  Stool consistency measured by the Bristol scale from 1(severe constipation) to 7 (severe diarrhea)
Patient-reported outcomes obtained from the bowel habit diary. | Each patient fills out the diary every day for one week at baseline, for one week starting at each day of the two interventions and for one week at the long term follow-up at week 26
  Median number of bowel openings per 24 hours.
Patient-reported outcomes obtained from the bowel habit diary. | Each patient fills out the diary every day for one week at baseline, for one week starting at each day of the two interventions and for one week at the long term follow-up at week 26
  Number of nightly bowel openings (from bedtime until morning).
Patient-reported outcomes obtained from the bowel habit diary. | Each patient fills out the diary every day for one week at baseline, for one week starting at each day of the two interventions and for one week at the long term follow-up at week 26
  Number of episodes with involuntary defaecation.
Patient-reported outcomes obtained from the bowel habit diary. | Each patient fills out the diary every day for one week at baseline, for one week starting at each day of the two interventions and for one week at the long term follow-up at week 26
  Glycemic control measured by patient reported use of insulin (IE).
Patient-reported measures from the schedule of side effects and telephone call 1 week after each intervention. | One week after each intervention
  Mild adverse events (grade 1) following FMT or placebo assessed by CTCAE v5.0.
Patient-reported outcomes from questionnaires. | at baseline and 4 weeks after each intervention period and at long term follow-up at week 26
  Change in Gastrointestinal syndrome rating scale - irritable bowel version questionnaire (GSRS-IBS)
Patient-reported outcomes from questionnaires. | at baseline and 4 weeks after each intervention period and at long term follow-up at week 26
  Change in patient assessment of upper gastrointestinal symptom severity index (PAGI-SYM)
Patient-reported outcomes from questionnaires. | at baseline and 4 weeks after each intervention period and at long term follow-up at week 26
  Change in irritable bowel syndrome impact scale (IBS-IS)
Objective measures from the wireless motility capsule. | at baseline and 4 weeks after each intervention period
  Transit time through the small intestine.
Objective measures from the wireless motility capsule. | at baseline and 4 weeks after each intervention period
  Colonic transit time.
Objective measures from the wireless motility capsule. | at baseline and 4 weeks after each intervention period
  pH drop from the small intestine to the colon.
Objective measures from the low-dose CT scan. | at baseline and 4 weeks after the first intervention
  Volume of the a) small intestine and b) the colon. Volume of gas in a) the small intestine and b) the colon.
Objective measures from the breath test. | at baseline and 4 weeks after the first intervention
  Rise in hydrogen PPM measured in breath test for small intestinal bacterial overgrowth.
Microbiota analysis on faecal samples. | at baseline and 4 weeks after each intervention period
  Alpha-diversity of faecal microbiota, 16S. Dysbiosis index.
Microbiota analysis on faecal samples. | at baseline and 4 weeks after each intervention period
  Dysbiosis index.
Blood samples. | at baseline and 4 weeks after each intervention period
  Glycemic control measured by HbA1C levels.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Krogh, MD, DMSc, PhD, Professor, Principal Investigator — Department of Hepatology and Gastroenterology, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jorgensen SMD, Hansen MM, Erikstrup C, Dahlerup JF, Hvas CL. Faecal microbiota transplantation: establishment of a clinical application framework. Eur J Gastroenterol Hepatol. 2017 Nov;29(11):e36-e45. doi: 10.1097/MEG.0000000000000958. PMID 28863010
- [Derived] Hoyer KL, Kornum DS, Baunwall SMD, Klinge MW, Drewes AM, Yderstraede KB, Mikkelsen S, Erikstrup C, Krogh K, Hvas CL. Repeated faecal microbiota transplantation for individuals with type 1 diabetes and gastroenteropathy. Diabetologia. 2025 Dec;68(12):2795-2806. doi: 10.1007/s00125-025-06544-x. Epub 2025 Sep 18. PMID 40965701
- [Derived] Hoyer KL, Dahl Baunwall SM, Kornum DS, Klinge MW, Drewes AM, Yderstraede KB, Thingholm LB, Mortensen MS, Mikkelsen S, Erikstrup C, Hvas CL, Krogh K. Faecal microbiota transplantation for patients with diabetes type 1 and severe gastrointestinal neuropathy (FADIGAS): a randomised, double-blinded, placebo-controlled trial. EClinicalMedicine. 2024 Dec 16;79:103000. doi: 10.1016/j.eclinm.2024.103000. eCollection 2025 Jan. PMID 39791110